CLINICAL TRIAL: NCT00168415
Title: A Study Using Botulinum Toxin Type A in Adolescents With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-075
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A

ARMS (1):
- 1 (Experimental): Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — 100 U up to 6 times during the study depending on the response to treatment
  Other Names: BOTOX®

SUMMARY:
A study using Botulinum Toxin Type A in adolescents with axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Marked axillary hyperhidrosis

Exclusion Criteria:

* Previous use of botulinum toxin for hyperhidrosis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2005-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Subject's assessment of the severity of hyperhidrosis using the HDS Scale | Monthly

SECONDARY OUTCOMES:
Measurement of axillary sweat production | Week 4, Week 8 and any re-injection visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Portland, Oregon, United States
- Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Glaser DA, Pariser DM, Hebert AA, Landells I, Somogyi C, Weng E, Brin MF, Beddingfield F. A Prospective, Nonrandomized, Open-Label Study of the Efficacy and Safety of OnabotulinumtoxinA in Adolescents with Primary Axillary Hyperhidrosis. Pediatr Dermatol. 2015 Sep-Oct;32(5):609-17. doi: 10.1111/pde.12620. Epub 2015 Jun 8. PMID 26059781